CLINICAL TRIAL: NCT02969083
Title: Neo-adjuvant Versus Adjuvant Chemotherapy in Upper Tract Urothelial Carcinoma: A Feasibility Phase II Randomized Clinical Trial ("URANUS")"
Brief Title: Feasibility of Neo-adjuvant Versus Adjuvant Chemotherapy in Upper Tract Urothelial Carcinoma
Acronym: URANUS
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The European Uro-Oncology Group (Other)
Collaborators: Centre for Human Drug Research, Netherlands (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: EudraCT 2016-004017-27
Record Dates: First submitted 2016-11-11; First posted 2016-11-21 (Estimated); Last update posted 2023-12-18 (Actual); Status verified 2023-03

CONDITIONS: Upper Tract Urothelial Carcinoma
Keywords: UTUC; Upper Tract Urothelial Carcinoma; Neoadjuvant chemotherapy; Adjuvant chemotherapy; Radical nephroureterectomy
MeSH Terms: interventions — Gemcitabine; Cisplatin; M-VAC protocol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Radical nephro-ureterectomy (RNU) (Other): Patients who dont fulfil inclusion criteria for chemotherapy treatment randomization (poor renal function: Glomerular Filtration Rate (GFR) <55 ml/min or unfit for cisplatin-based chemotherapy)
  Interventions: Procedure: RNU
- Gemcitabine/Cisplatin plus RNU (Other): Patients who fulfil inclusion criteria for cisplatinum-based chemotherapy (renal function: GRF > or = 55 ml/min) receiving 3 cycles of Gemcitabine (1000 mg/m2) + Cisplatin (70 mg/m2) every 3 weeks before surgery
  Interventions: Procedure: RNU; Drug: Gemcitabine/Cisplatin
- RNU plus Gemcitabine/Cisplatin (Other): Patients who fulfil inclusion criteria for cisplatinum-based chemotherapy (renal function: GRF > or = 55 ml/min) receiving 3 cycles of Gemcitabine (1000 mg/m2) + Cisplatin (70 mg/m2) every 3 weeks after surgery
  Interventions: Procedure: RNU; Drug: Gemcitabine/Cisplatin
- M-VAC protocol plus RNU (Other): Patients who fulfil inclusion criteria for cisplatinum-based chemotherapy (renal function: GRF > or = 55 ml/min) receiving 3 cycles of MVAC every 2 weeks (Methotrexate (30 mg /m²) , Vinblastine (3 mg /m²) , Adriamycin (30 mg /m²) , and Cisplatin (70 mg /m²) before surgery
  Interventions: Procedure: RNU; Drug: M-VAC Protocol
- RNU plus M-VAC protocol (Other): Patients who fulfil inclusion criteria for cisplatinum-based chemotherapy (renal function: GRF > or = 55 ml/min) receiving 3 cycles of MVAC every 2 weeks (Methotrexate (30 mg /m²) , Vinblastine (3 mg /m²) , Adriamycin (30 mg /m²) , and Cisplatin (70 mg /m²) after surgery
  Interventions: Procedure: RNU; Drug: M-VAC Protocol

INTERVENTIONS:
Procedure: RNU — Radical surgical removal by open or laparoscopic access
  Other Names: Radical nephro-ureterectomy
Drug: Gemcitabine/Cisplatin — Gemcitabine (1000 mg/m²) day 1 and 8 and Cisplatin (70 mg/m²) day 1
  Other Names: Gemcitabine plus Cisplatin
  Arms: Gemcitabine/Cisplatin plus RNU; RNU plus Gemcitabine/Cisplatin
Drug: M-VAC Protocol — Methotrexate (30 mg /m²) and Vinblastine 3 (mg /m²) day 1; Adriamycin 30 mg /m² and Cisplatin 70 mg /m² in day2
  Other Names: DD MVAC
  Arms: M-VAC protocol plus RNU; RNU plus M-VAC protocol

SUMMARY:
The aim of this study is to explore feasibility of Upper Tract Urothelial Carcinoma (UTUC) treatments based in real world data in various European countries. The study will allow to gain insight in the true proportion of patients that fit to receive complete cisplatin-based neo-adjuvant or adjuvant chemotherapy, and the proportion and clinical outcome of patients with poor prognostic factors (PS and renal function) who receive only standard treatment (Radical nephroureterectomy (RNU)). This comparison will be made using a uniform diagnostic and treatment protocol.

DETAILED DESCRIPTION:
There are no definitive treatment recommendations for patients diagnosed with UTUC. Radical nephroureterectomy (RNU) has been considered the gold standard treatment for UTUC. However due to the high recurrence rates reported, patients are often offered perioperative chemotherapy provided that they have a good renal function and performance status. With regard to the choice of chemotherapy treatment, there are also no clear recommendations since there are no data from randomized studies. If perioperative chemotherapy is considered in daily practice, gemcitabine/cisplatin regimen is often chosen and occasionally dd-MVAC.

The aim of this study is to explore feasibility of UTUC treatments based in real world data in various European countries. Patients who fulfil good prognostic factors (inclusion criteria for treatment randomization) will be allocated to neo-adjuvant (Arm B) or adjuvant (Arm C) chemotherapy (receiving 3 cycles of gemcitabine/cisplatin or dose dense Methotrexate, Vinblastine, Adriamycin, and Cisplatin (MVAC). Patients who don't fulfil criteria for treatment randomization will undergo Radical nephroureterectomy (RNU) only (Arm A). Patients will be followed up for 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Age > 18 years
* Histological and radiological defined UTUC: Histologically-confirmed diagnosis of predominantly urothelial carcinoma of the upper urinary tract Patients with UTUC cT2-pT4 cN0-N1 M0 (TNM classification)
* Women with negative serum pregnancy test within 14 days of first dose of study treatment and agreement to use effective contraception
* Patients without bladder cancer or with concomitant non muscle invasive bladder cancer
* Adequate organ system function defined as follows: Hematologic: Absolute neutrophil count (ANC) 1.5 X 109/L; Haemoglobin 5.6 mmol/L (9.02g/dL); Platelets 100 X 109/L; Prothrombin time (PT) or international normalized ratio (INR)b 1.2 X ULN; Activated partial thromboplastin time (aPTT)1.2 X Upper limit of normal (ULN). Hepatic: Total bilirubin 1.5 X ULN; Alanine amino transferase (ALT) and Aspartate aminotransferase (AST) 2.5 X ULN. Renal: GRF <or> 55 ml/min: Electrolytes: potassium and calcium: within normal limits.
* CT scan of the chest, abdomen and pelvis and Bone scan without evidence of distant metastasis

Exclusion Criteria:

* Histology of pure adenocarcinoma, pure squamous cell carcinoma, sarcomatoid or predominant small cell carcinoma.
* History of cardiovascular conditions within the past 6 months.
* Incidentally found asymptomatic pulmonary embolism (PE) or recent deep vein thrombosis (DVT) is not an exclusion criteria but requires anticoagulation treatment.
* Any major contraindication to a surgical procedure.
* Any serious and/or unstable pre-existing medical, psychiatric, or other condition that could interfere with subject's safety, provision of informed consent, or compliance to study procedures.
* Active infection contraindicating chemotherapy
* Other active neoplasms. Patients with in situ cervical carcinoma, non-melanoma skin cancer or prostate cancer T1 Gleason <7, Prostate specific antigen (PSA) <10. Patients with past medical history of cancer can be included if diagnosed at least 4 years ago.
* Concomitant muscle invasive bladder cancer
* Patients who have been or still are on methotrexate treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2018-05-28 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Proportion of UTUC patients randomized to neo- or adjuvant chemotherapy that is actually able to start and finalize three courses of planned chemotherapy | 6 months
  Percentage of patients randomised to adjuvant or neo-adjuvant treatment

SECONDARY OUTCOMES:
Disease Free Survival (DFS) | 1-2 years
  time from randomisation to local recurrence or distant metastasis
Overall Survival (OS) | 1-2 years
  time from randomisation to death for any cause different from urothelial carcinoma
Cancer-Specific Survival (CSS) | 1-2 years
  time from randomisation to death from urothelial carcinoma

CONTACTS AND LOCATIONS:
Overall Officials: Susanne Osanto, MD, PhD, Principal Investigator — Leiden University Medical Centre
Locations (29):
- Netherlands (4):
  - Radboud University Medical Centre, Nijmegen, Gelderland
  - Leiden University Medical Centre, Leiden, South Holland
  - Alrijne Ziekenhuis, Leiderdorp, South Holland
  - Canisius Wilhelmina Ziekenhuis, Nijmegen
- Haukeland University Hospital, Bergen, Norway
- Spain (24):
  - Complejo Hospitalario Universitario A Coruña, A Coruña
  - Hospital Universitario German Trias i Pujol, Badalona
  - Fundacion Puigvert, Barcelona
  - Hospital Clinico de Barcelona, Barcelona
  - Hospital San Pau, Barcelona
  - Hospital Universitario Vall d'Hebron, Barcelona
  - Hospital Universitario de Basurto, Bilbao
  - Hospital Universitari de Girona Doctor Josep Trueta, Girona
  - Hospital Universitario Clínico San Cecilio, Granada
  - Hospital de Jerez, Jerez de la Frontera
  - Hospital Complex Insular-Materno Infantil, Las Palmas
  - Clinica Universitaria de Navarra, Madrid
  - Fundacion Jimenez Diaz, Madrid
  - Hospital ramón y Cajal, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Clinico Universitario Virgen de la Arrixaca, Murcia
  - Hospital General Universitario Morales Meseguer, Murcia
  - Complejo Hospitalario de Navarra, Pamplona
  - Hospital Parc Taulí, Sabadell
  - Hospital Universitario de Salamanca, Salamanca
  - Hospital Universitario Marques de Valdecilla, Santander
  - Hospital Virgen del Rocio, Seville
  - Fundacion Instituto Valenciano de Oncologia, Valencia
  - Hospital Clinico Universitario Lozano Blesa, Zaragoza

IPD SHARING:
Plan to Share IPD: No
The results obtained in this study will be disseminated and published

REFERENCES:
- [Derived] Hird AE, Magee DE, Cheung DC, Sander B, Sridhar S, Nam RK, Kulkarni GS. Neoadjuvant Versus Adjuvant Chemotherapy for Upper Tract Urothelial Carcinoma: A Microsimulation Model. Clin Genitourin Cancer. 2021 Apr;19(2):e135-e147. doi: 10.1016/j.clgc.2020.10.001. Epub 2020 Oct 13. PMID 33168398